CLINICAL TRIAL: NCT06943599
Title: Village Integrated Eye Worker II Linkage-to-Care Trial
Brief Title: Strategies for Improving Linkage-to-Care After Eye Disease Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Seva Foundation (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-22776-3; UG1EY036346 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Age Related Macular Degeneration; Diabetic Retinopathy; Glaucoma
Keywords: Eye Diseases; mass screening; patient compliance; retention in care
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Glaucoma; Eye Diseases; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text Message Reminders (Experimental)
  Interventions: Other: Text Message Reminder
- Health Worker (Experimental)
  Interventions: Other: Health Worker Visit
- No Intervention (No Intervention)

INTERVENTIONS:
Other: Text Message Reminder — Participants referred to the eye hospital after screening will receive a text message reminding them to attend their referral visit.
  Arms: Text Message Reminders
Other: Health Worker Visit — Participants referred to the eye hospital after screening will receive a home visit from a health worker reminding them to attend their referral visit.
  Arms: Health Worker

SUMMARY:
The goal of this randomized, parallel-group, controlled trial is to compare methods of improving linkage-to-care for participants in the Village Integrated Eye Worker II (VIEW II) trial who are referred to the eye hospital following eye disease screening. Participants who are referred to the hospital at an eye screening visit will be randomized to three different linkage-to-care interventions: (1) text message reminders, (2) reminders from health workers, or (3) no intervention. The primary outcome of the trial will be whether or not the participant presented to the eye hospital for a referral visit by 21 days following screening.

ELIGIBILITY:
Inclusion Criteria:

- Participant of the VIEW II study referred to the eye hospital at their eye screening visit.

Exclusion Criteria:

* Residence in an area without reliable mobile connectivity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Referral Visit Attendance | 21 days after screening
  The count of participants who attend the referral visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Keenan, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including age, cluster identifier, referral visit attendance
Supporting Information: Study Protocol
Time Frame: De-identified data will be shared after publication of the major findings of the study, which we anticipate will occur around 6 months after the study conclusion.
Access Criteria: Other investigators can access the data if approved by the Trial Coordinating Center. Requests should be sent to the study contact(s).
URL: https://osf.io/fgvrt/